CLINICAL TRIAL: NCT03739255
Title: Treatment of Postoperative Discomfort/Pain and Facilitation of Corneal Reepithelialization After Photorefractive Keratectomy
Brief Title: Facilitation of Corneal Re-epithelialization After Photorefractive Keratectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SynsLaser Kirurgi AS (Other)
Collaborators: Laboratoires Thea (Industry)
Responsible Party: Principal Investigator, Aleksandar Stojanovic, Medical Director, SynsLaser Kirurgi AS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/1985/REK sør-øst
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Corneal Erosion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cacicol20 (Experimental): One drop of Cacicol20 will be applied 4-6 hours after the surgery, in one of the randomly chosen eye, and thereafter one drop daily until the reepithelialization is completed.
  Interventions: Device: Cacicol20
- Placebo (Placebo Comparator): One drop of conservative free artificial tear (Oculac, Thea Laboratories) will be applied to one eye at the same time when Cacicol20 is instilled to the other eye.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Cacicol20 — Cacicol20 is supplied as a sterile single-dose solution of alpha 1-6 poly-carboxymethyl glucose sulfate One drop is instilled at each application to impregnate cornea.
  Other Names: regenerative medicine
  Arms: Cacicol20
Device: Placebo — Ocluac is artificial tear which contains Hydroxypropylmethyl Cellulose and Sodium Chloride, It is presented in a 0.4 mL vial. One drop is delivered at each application.
  Arms: Placebo

SUMMARY:
Photorefractive keratectomy (PRK) or surface ablation is one of the most commonly used surgical procedures to correct refractive errors, which was proved to be safe and effective. In PRK, the corneal epithelium is removed by various techniques such as diluted alcohol, manual debridement, brush, or excimer laser, before the refractive excimer laser ablation of the corneal stroma. Compared to laser in situ keratomileusis (LASIK), the two main drawbacks for PRK are slower visual recovery and discomfort in the immediate postoperative period, due to the epithelial removal.

Corneal healing is a complex process involving cellular interaction and reaction with various molecules (proteases, growth factors, and epithelial and stromal cytokines). Enhanced corneal re-epithelialization may reduce the risk for corneal infection and stromal scarring or melting. Over the past few years, a new type of matrix therapy by ReGeneraTing Agent (RGTA) has provided encouraging results, accelerating the healing of chronic skin ulcers in diabetes or vascular origin. RGTAs mimic the action of heparin sulfate molecules, breaking the negative repair-destruction cycle occurring in chronic lesions and inhibit proteolytic enzymes in vitro. In the domain of ophthalmology, RGTA has been reported to show encouraging results in the treatment of corneal ulcer and dystrophies of various etiologies.

The Cacicol20 is an RGTA that binds to matrix proteins to protect them from proteolysis; the extracellular matrix microenvironment protection improves the production of signals and growth factors needed for tissue healing. It is supplied as a sterile single-dose solution of alpha 1-6 poly-carboxymethyl glucose sulfate described and synthesized as in US Patent Number 6689741, with dextran T40 and 0.9% sodium chloride as excipients. It contains no component of animal or biological origin, and penetrates into the cornea without crossing Descemet´s membrane (no intraocular penetration). The Cacicol20 has been reported to be effective in treatment of neurotrophic ulcers and persistent epithelial defects which were unresponsive to the common treatment approaches. Therefore, we expect that the Cacicol20 may facilitate the corneal re-epithelialization after PRK.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bilateral PRK surgeries for treatment of refractive error
* Age over 18 years
* Refractive stability for at least 2 years

Exclusion Criteria:

* Ocular pathology, including keratoconus or suspected keratoconus, glaucoma, and epithelial defects
* Previous corneal surgery
* Systemic disease that might affect corneal wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Re-epithelialization time | 5 days postoperatively
  The patients will be examined daily the changes of reepithelialization area, until the re-epithelialization is complete. The days that takes for complete reepithelialization will be recorded.

SECONDARY OUTCOMES:
Discomfort during reepithelialization | 5 days postoperatively
  Patient´s subjective evaluation of ocular symptoms including pain, burning, stinging, tearing, and photophobia in the two eyes, with score ranging from 0-5 (0 representing absence of symptom and 5 representing unbearable symptom) will be performed daily

OTHER OUTCOMES:
Postoperative corneal epithelial thickness | 1 week and 1 month postoperatively
  Epithelial thickness in the central 2 mm and mid-peripheral (2-5 mm) cornea will be measured in µm using anterior segment spectrum-domain optical coherence tomography
Inflammatory cytokine | Preoperatively, 24 hours and 72 hours after the surgery
  Concentration of inflammatory cytokines in tears including interleukin 1ß (IL-1ß), IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17A, IL-1RA (receptor antagonist), eotaxin, basic fibroblast growth factor (bFGF/FGF2), granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF), interferon gamma (IFN-γ), interferon gamma-induced protein 10 (IP-10), monocyte chemoattractant protein 1 (MCP-1), macrophage inflammatory protein 1α (MIP-1α/CCL3), MIP-1B, platelet-derived growth factor bb (PDGF-BB), regulated-on-activation normal T cell expressed and secreted (RANTES), tumor necrosis factor alpha (TNF-α), and vascular endothelial growth factor (VEGF) will be measured using Multiplex analysis
Postoperative uncorrected visual acuity | 1 week, 1 month postoperatively
  Uncorrected visual acuity will be measured using Snellen visual acuity chart
Refractive outcome | 1 month and 3 months postoperatively
  Subjective manifest refraction will be performed and spherical equivalent (SE) will be recorded in diopters
Protein expression in tear fluid | Preoperatively, 24 hours and 72 hours after the surgery
  The proteome of tear fluid will be examined through Liquid chromatographymass spectrometry (LC-MS)
Postoperative complications | 1 month and 3 months postoperatively
  The incidence of postoperative complications (infection, haze formation, delayed epithelial healing) will be recorded in percentage
Postoperative dry eye disease severity level | 1 month and 3 months postoperatively
  Clinical dry eye tests including ocular surface disease index (OSDI) questionnaire (score between 0-100, whith higher values presenting more severe dry eye symptoms), tear break-up time (recorded in seconds), ocular surface staining recorded using Oxford scale (0-15, with higher value representing more ocular surface staining), which will be used to determine the dry eye severity level, according to the 2007 Dry Eye Workshop (DEWS) report

REFERENCES:
- [Result] Groah SL, Libin A, Spungen M, Nguyen KL, Woods E, Nabili M, Ramella-Roman J, Barritault D. Regenerating matrix-based therapy for chronic wound healing: a prospective within-subject pilot study. Int Wound J. 2011 Feb;8(1):85-95. doi: 10.1111/j.1742-481X.2010.00748.x. Epub 2010 Nov 16. PMID 21078132
- [Result] Garcia-Filipe S, Barbier-Chassefiere V, Alexakis C, Huet E, Ledoux D, Kerros ME, Petit E, Barritault D, Caruelle JP, Kern P. RGTA OTR4120, a heparan sulfate mimetic, is a possible long-term active agent to heal burned skin. J Biomed Mater Res A. 2007 Jan;80(1):75-84. doi: 10.1002/jbm.a.30874. PMID 16958049
- [Result] Aifa A, Gueudry J, Portmann A, Delcampe A, Muraine M. Topical treatment with a new matrix therapy agent (RGTA) for the treatment of corneal neurotrophic ulcers. Invest Ophthalmol Vis Sci. 2012 Dec 13;53(13):8181-5. doi: 10.1167/iovs.12-10476. PMID 23150626
- [Result] Kymionis GD, Liakopoulos DA, Grentzelos MA, Diakonis VF, Klados NE, Tsoulnaras KI, Tsilimbaris MK, Pallikaris IG. Combined topical application of a regenerative agent with a bandage contact lens for the treatment of persistent epithelial defects. Cornea. 2014 Aug;33(8):868-72. doi: 10.1097/ICO.0000000000000169. PMID 24937169